CLINICAL TRIAL: NCT02090803
Title: Assessment of Human Herpes Virus Reactivation 6 Post Autologous Stem Cells , Prospective, Open, Multicenter Study
Brief Title: Assessment of Human Herpes Virus Reactivation 6 Post Autologous Stem Cells
Acronym: VIRAUTO6
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-01; 2012-A000243-40 (Other: Agence Nationale de Sécurité du Médicament)
Record Dates: First submitted 2014-03-17; First posted 2014-03-18 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2014-03

CONDITIONS: Hematologic Diseases
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Graft of autologous hematopoietic stem cells

SUMMARY:
The purpose of this study is to assess the human herpes virus reactivation 6 post autologous stem cells in 196 patients. The aim of our study was to describe the incidence of reactivation of HHV-6 in patients requiring autologous HSCT and determine the pathogenic role in this target population.

ELIGIBILITY:
Inclusion Criteria:

* all patients hospitalized in the Hematology Clinic of Saint-Etienne and Clermont-Ferrand and receiving autologous hematopoietic stem cells, according to the decision of the Consultative Meeting Multidisciplinary service;
* Autologous recipients are included irrespective of causal hemopathy (myeloma, lymphoma, acute leukemia, mainly).

Exclusion Criteria:

* The non-consenting patients or unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patient
Sampling Method: Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2012-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
HHV-6 biological reactivation | 40 days
  HHV-6 biological reactivation (blood viral load) is defined by a detectable viral load HHV-6 and> 450 copies / mL on two occasions one week apart.

SECONDARY OUTCOMES:
Aplasia output or engraftment | 40 days
Reconstitution of hematopoiesis | 40 days
Disease HHV-6 | 40 days

CONTACTS AND LOCATIONS:
Overall Officials: Marie Balsat, MD, Study Chair — Institut de Cancérologie Lucien Neuwirth
Locations (3):
- France (3):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - HCL, Lyon
  - CHU Saint-Etienne - laboratoire de virologie, Saint-Etienne

REFERENCES:
- [Background] De Bolle L, Naesens L, De Clercq E. Update on human herpesvirus 6 biology, clinical features, and therapy. Clin Microbiol Rev. 2005 Jan;18(1):217-45. doi: 10.1128/CMR.18.1.217-245.2005. PMID 15653828
- [Background] Boutolleau D, Duros C, Bonnafous P, Caiola D, Karras A, Castro ND, Ouachee M, Narcy P, Gueudin M, Agut H, Gautheret-Dejean A. Identification of human herpesvirus 6 variants A and B by primer-specific real-time PCR may help to revisit their respective role in pathology. J Clin Virol. 2006 Mar;35(3):257-63. doi: 10.1016/j.jcv.2005.08.002. Epub 2005 Sep 23. PMID 16183328
- [Background] Yamanishi K, Okuno T, Shiraki K, Takahashi M, Kondo T, Asano Y, Kurata T. Identification of human herpesvirus-6 as a causal agent for exanthem subitum. Lancet. 1988 May 14;1(8594):1065-7. doi: 10.1016/s0140-6736(88)91893-4. PMID 2896909
- [Background] Santoro F, Kennedy PE, Locatelli G, Malnati MS, Berger EA, Lusso P. CD46 is a cellular receptor for human herpesvirus 6. Cell. 1999 Dec 23;99(7):817-27. doi: 10.1016/s0092-8674(00)81678-5. PMID 10619434
- [Background] Agut H. Deciphering the clinical impact of acute human herpesvirus 6 (HHV-6) infections. J Clin Virol. 2011 Nov;52(3):164-71. doi: 10.1016/j.jcv.2011.06.008. Epub 2011 Jul 22. PMID 21782505
- [Background] Ljungman P, Wang FZ, Clark DA, Emery VC, Remberger M, Ringden O, Linde A. High levels of human herpesvirus 6 DNA in peripheral blood leucocytes are correlated to platelet engraftment and disease in allogeneic stem cell transplant patients. Br J Haematol. 2000 Dec;111(3):774-81. PMID 11122137
- [Background] Ljungman P. Immune reconstitution and viral infections after stem cell transplantation. Bone Marrow Transplant. 1998 Apr;21 Suppl 2:S72-4. PMID 9630332
- [Background] Agut H. [Acute human herpesvirus 6 (HHV-6) infections: when and how to treat?]. Pathol Biol (Paris). 2011 Apr;59(2):108-12. doi: 10.1016/j.patbio.2010.07.015. Epub 2010 Sep 15. French. PMID 20832191
- [Background] Kamble RT, Clark DA, Leong HN, Heslop HE, Brenner MK, Carrum G. Transmission of integrated human herpesvirus-6 in allogeneic hematopoietic stem cell transplantation. Bone Marrow Transplant. 2007 Sep;40(6):563-6. doi: 10.1038/sj.bmt.1705780. Epub 2007 Jul 16. PMID 17637686
- [Background] Lee SO, Brown RA, Razonable RR. Clinical significance of pretransplant chromosomally integrated human herpesvirus-6 in liver transplant recipients. Transplantation. 2011 Jul 27;92(2):224-9. doi: 10.1097/TP.0b013e318222444a. PMID 21629177
- [Background] Moreau P, Facon T, Attal M, Hulin C, Michallet M, Maloisel F, Sotto JJ, Guilhot F, Marit G, Doyen C, Jaubert J, Fuzibet JG, Francois S, Benboubker L, Monconduit M, Voillat L, Macro M, Berthou C, Dorvaux V, Pignon B, Rio B, Matthes T, Casassus P, Caillot D, Najman N, Grosbois B, Bataille R, Harousseau JL; Intergroupe Francophone du Myelome. Comparison of 200 mg/m(2) melphalan and 8 Gy total body irradiation plus 140 mg/m(2) melphalan as conditioning regimens for peripheral blood stem cell transplantation in patients with newly diagnosed multiple myeloma: final analysis of the Intergroupe Francophone du Myelome 9502 randomized trial. Blood. 2002 Feb 1;99(3):731-5. doi: 10.1182/blood.v99.3.731. PMID 11806971
- [Background] Leong HN, Tuke PW, Tedder RS, Khanom AB, Eglin RP, Atkinson CE, Ward KN, Griffiths PD, Clark DA. The prevalence of chromosomally integrated human herpesvirus 6 genomes in the blood of UK blood donors. J Med Virol. 2007 Jan;79(1):45-51. doi: 10.1002/jmv.20760. PMID 17133548
- [Background] Ogata M. Human herpesvirus 6 in hematological malignancies. J Clin Exp Hematop. 2009 Nov;49(2):57-67. doi: 10.3960/jslrt.49.57. PMID 19907110